CLINICAL TRIAL: NCT05352763
Title: An Open-Label Extension of the PTI-125-04 Study Evaluating the Safety and Long-Term Treatment of Simufilam in Mild-to-Moderate Alzheimer's Disease Patients
Brief Title: Open-Label Extension of the PTI-125-04 Study in Mild-to-Moderate Alzheimer's Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Cassava Sciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTI-125-09
Record Dates: First submitted 2022-04-04; First posted 2022-04-29 (Actual); Results first posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-07

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Simufilam

STUDY DESIGN:
Intervention Model Description: Open-label extension study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Simufilam 100 mg (Experimental): simufilam 100 mg oral tablets, b.i.d.
  Interventions: Drug: simufilam

INTERVENTIONS:
Drug: simufilam — simufilam 100 mg oral tablet, twice daily
  Other Names: PTI-125

SUMMARY:
This is a 96-week extension study of open-label simufilam 100 mg b.i.d. for mild-to-moderate Alzheimer's disease subjects who completed the Phase 2 study, PTI-125-04. The study will evaluate safety and long-term treatment. Safety will be assessed by AE monitoring, clinical labs, urinalysis, vital signs, ECGs, and C-SSRS.

DETAILED DESCRIPTION:
This is an open-label 96-week extension study of open-label simufilam 100 mg b.i.d. for subjects who completed the Phase 2 study, PTI-125-04. All subjects will provide consent to enroll into this study. Simufilam will be administered as coated oral tablets. The last study visit, Month 24, from the PTI-125-04 study will be used for the Study Day 1 visit assessments in this extension study. Clinic visits will occur every 12 weeks ±10 days. A complete physical examination will be performed at Study Day 1, Week 48 and Week 96. Subjects will return to the clinic every 12 weeks for safety assessments of vital signs, AE monitoring, C-SSRS, and drug dispensation and accountability. Blood draws for clinical laboratory testing, urine collection for urinalysis, and ECGs will be performed at Study Day 1 and Weeks 24, 48, 72, and 96. Safety will be evaluated by adverse event monitoring, vital signs, clinical labs, and the Columbia Suicide Severity Rating Scale (C-SSRS).

ELIGIBILITY:
1. Must have completed the PTI-125-04 study or Week 96 in the PTI-125-09 study.
2. Male subjects must be willing to continue use of contraception during the study. With female partners of childbearing potential, male subjects, regardless of their fertility status, must agree to either remain abstinent or use condoms in combination with one additional highly effective method of contraception (e.g., oral or implanted contraceptives, or intrauterine devices) or an effective method of contraception (e.g., diaphragms with spermicide or cervical sponges) during the study and for 14 days after study drug dosing has been completed.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-05-12 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chris Cook, JD, Study Chair — Chief Operating and Legal Officer
Locations (11):
- United States (9):
  - Cognitive Clinical Trials, Gilbert, Arizona
  - Valley Research Center, Inc., Imperial, California
  - Brain Matters Research, Delray Beach, Florida
  - Neuropsychiatric Research Center of Southwest Florida, Fort Myers, Florida
  - IMIC Research, Palmetto Bay, Florida
  - Cognitive Clinical Trials, Papillion, Nebraska
  - Advanced Memory Research Institute of NJ, Toms River, New Jersey
  - the Ohio State University, Columbus, Ohio
  - Senior Adults Specialty Research, Austin, Texas
- Canada (2):
  - Recherches Neuro-Hippocampe Inc., d/b/a Ottawa Memory Clinic, Ottawa, Ontario
  - Toronto Memory Program ULC, Toronto, Ontario

RESULTS

PARTICIPANT FLOW:
Groups:
- Simufilam 100 mg: simufilam 100 mg oral tablet, twice daily
  simufilam: simufilam 100 mg oral tablets
Period: Overall Study
Arm/Group | Simufilam 100 mg
Started | 90
Completed | 21
Not Completed | 69

BASELINE CHARACTERISTICS:
Arm/Group | Simufilam 100 mg
Number analyzed (Participants) | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 71
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.2 (8.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55
  Male | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 83
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 87
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Adverse Event Monitoring
Description: Number of Participants with Adverse Events
Time Frame: Baseline to 96 Weeks
Population: Safety Analysis Population
Measure: Count of Participants; unit: Participants
Groups:
- Simufilam 100 mg: simufilam 100 mg oral tablet, twice daily
  simufilam: simufilam 100 mg oral tablet, twice daily
Arm/Group | Simufilam 100 mg
Number analyzed (Participants) | 90
Participants | 90
Statistical Analysis 1: Comparison: Simufilam 100 mg; Test type: Other — No statistical analysis performed; The classical summary of count and percentages will be provided for basic safety tabulations and dispositions as appropriate. All data will be presented in by-subject data listings. No inferential statistics will be produced

ADVERSE EVENTS:
Time Frame: Up to 2 years
Groups:
- Simufilam 100 mg: simufilam 100 mg oral tablets, b.i.d.
  simufilam: simufilam 100 mg oral tablets
Arm/Group | Simufilam 100 mg
All-Cause Mortality (participants affected / at risk) | 0/90
Serious Adverse Events (participants affected / at risk) | 15/90
Other Adverse Events (participants affected / at risk) | 43/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Simufilam 100 mg (N=90)
Atrial fibrillation (Cardiac disorders) | 1
Abdominal hernia perforation (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Pelvic mass (Gastrointestinal disorders) | 1
Sepsis (Infections and infestations) | 1
COVID-19 (Infections and infestations) | 2
Cellulitis (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Rib fracture (Injury, poisoning and procedural complications) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 2
Agitation (Psychiatric disorders) | 1
Immobile (Social circumstances) | 1
Deep vein thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Simufilam 100 mg (N=90)
Urinary tract infection (Infections and infestations) | 15
Fall (Injury, poisoning and procedural complications) | 14
COVID-19 (Infections and infestations) | 10
Anxiety (Psychiatric disorders) | 8
Upper respiratory tract infection (Infections and infestations) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2024-09-18): https://cdn.clinicaltrials.gov/large-docs/63/NCT05352763/Prot_000.pdf
  • Statistical Analysis Plan (2025-02-10): https://cdn.clinicaltrials.gov/large-docs/63/NCT05352763/SAP_001.pdf